CLINICAL TRIAL: NCT00533065
Title: Effects of the Cholinesterase Inhibitor Donepezil on Organic and Functional Deficits Associated With Age-Related Decrease of Growth Hormone
Brief Title: Effects of Donepezil on Deficits Associated With Age-Related Decrease of Growth Hormone
Acronym: GH-003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Karl Heinz Tragl MD, Ludwig Boltzmann Institute of Aging Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GH-003; EudraCT-Nr. 2005-001315-22; Ethics-commission: 05-052-0605
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Elderly
Keywords: Aging
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Donepezil — week1 - week12: 1 tablet per day (5mg) week13 - week52: 1 tablet per day (10mg)

SUMMARY:
The planned study has two purposes:

1. It is to provide evidence that the administration of a cholinesterase inhibitor will result in an increase of IGF-I (primary variable) and in an increase of the secretion growth hormone (secondary variable) that can be maintained throughout the treatment-period of one year.
2. The study also tests the hypothesis that maintenance of increased blood levels of growth hormone and IGF-I can stop or delay the age-related changes of body composition (secondary variables) .

ELIGIBILITY:
Inclusion Criteria:

* Aged between 70 and 80 years

Exclusion Criteria:

* Cardiac arrhythmias (sick sinus syndrome, AV block, sino-atrial block),
* Treatment with beta-blockers, NSAIDs or cholinergic agonists,
* Known hypersensitivity to donepezil hydrochloride, piperidine derivatives or to any excipients used in the formulation,
* Gastric and duodenal ulcer,
* Severe renal and hepatic impairment,
* Urinary congestion (prostatic hypertrophy),
* Obstructive pulmonary disease (bronchial asthma);

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Serum IGF1 | one year

SECONDARY OUTCOMES:
Growth hormone, body composition variables | one year

CONTACTS AND LOCATIONS:
Overall Officials: Karl H Tragl, MD, Study Director — Ludwig Boltzmann Institute of Aging Research
Locations (1):
- Ludwig Boltzmann Institute, Vienna, Vienna, Austria